CLINICAL TRIAL: NCT00930423
Title: Complement Activation During Hemodialysis in Atypical Hemolytic Uraemic Syndrome as Underlying Kidney Disease.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/270
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2014-12

CONDITIONS: Atypical Hemolytic Uraemic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cases: patients with endstage renal failure due to atypical uraemic syndrome treated with hemodialysis.
- controls: patiënts with endstage renal failure due to a non complement consuming nephropathy treated with hemodialysis.

SUMMARY:
Atypical hemolytic uraemic syndrome is caused by defects in the regulating factors in the alternative pathway of the complement system. Triggering can cause an uncontrolled complement activation with endothelial damage and thrombotic micro-angiopathy, especially in the kidneys. This can result in endstage renal failure. Complement activation during hemodialysis has been described as a result of contact between blood and the dialysis membrane. Our hypothesis is that patients with atypical hemolytic uraemic syndrome have a stronger complement activation during hemodialysis than patients with another underlying kidney disease. This could be a reason to treat patients with endstage renal failure due to atypical hemolytic uraemic syndrome preferentially with peritoneal dialysis instead of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* cases: endstage renal failure due to atypical hemolytic uraemic syndrome treated with hemodialysis.
* controls: endstage renal failure due to a non complement consuming nephropathy treated with hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with endstage renal failure treated in het University Hospital of Ghent
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
C3a-des-Arg measuring (as a marker of activation). | at time 0, at 15 minutes, at 60 minutes and at 180 minutes
white blood cell count | before and after 15 minutes of hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be